CLINICAL TRIAL: NCT06977243
Title: Effect of "Online MedEd" Intern Boot Camp Training on First Year Residents' Well-being: A Pilot Randomized Controlled Trial
Brief Title: Online MedEd Intern Bootcamp: Online Training for First Year Residents
Acronym: OME-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Raji Ayinla, Director of Medicine, New York City Health and Hospitals Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-08-130-273(HHC)
Record Dates: First submitted 2025-05-06; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Burnout Among First Year Residents
Keywords: Burnout; Wellness; Residents; Bootcamp
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Enrolled into a 7 weeks online training program from May 13 2025 to June 30 2025
  Interventions: Behavioral: Online MedEd Intern Bootcamp
- Control (No Intervention): The control group participants will receive residency orientation as per standard practice during June 2025, with no training sessions prior to starting the orientation to residency. The control group will be offered access to the online platform after completion of this study

INTERVENTIONS:
Behavioral: Online MedEd Intern Bootcamp — 7 weeks, online training program
  Arms: Intervention

SUMMARY:
This single-center, parallel-group randomized controlled trial will evaluate whether a seven-week, web-based "Online MedEd Intern Boot Camp" (OME-IB) program reduces burnout in incoming first-year residents at NYC Health + Hospitals/Harlem. Eligible participants are PGY-1 physicians starting in July 2025 in Internal Medicine, Pediatrics, Emergency Medicine, Surgery, Psychiatry, Infectious Disease, or Nephrology who have not previously completed U.S. postgraduate training. After consent and baseline surveys, approximately 26 interns will be randomized 1:1 (stratified by sex and specialty) to either (1) immediate access to the OME-IB platform plus 14 peer-facilitated, one-hour Zoom sessions on mental health, time management, documentation, and oral presentation over May-June 2025, or (2) usual residency orientation without Boot Camp access until study completion.

The primary outcome is mean Maslach Burnout Inventory-Emotional Exhaustion (MBI-EE) score six months into residency. Secondary outcomes at six months include mean Copenhagen Burnout Inventory personal-burnout subscale, Mini ReZ supportive-work-environment/work-pace/resident-experience subscales, and Patient Health Questionnaire-9 (PHQ-9) depression score. Surveys are administered via REDCap at baseline (pre-intervention), three months, and six months; analyses follow an intention-to-treat approach with linear mixed models. Qualitative interviews will explore participants' experiences four months into residency. Findings will inform refinement of the OME-IB curriculum and future multi-site trials aimed at improving resident well-being.

DETAILED DESCRIPTION:
Scientific Rationale: Burnout in early postgraduate physicians has been linked to elevated emotional-exhaustion scores, major medical errors, and a 370 % rise in suicidal ideation during the first three months of training. Guided by the Job-Demands/Resources framework, OME-IB is designed to enhance job control (time-management, documentation efficiency) and personal resources (peer support, resilience skills) to offset the high demands of residency. Prior pilot work with web-based cognitive-behavioral programs in interns has shown clinically meaningful reductions in depressive symptoms, but no randomized evidence exists for a comprehensive boot-camp format that couples asynchronous video content with live, peer-led skills practice.

Intervention Engineering and Fidelity

The OME-IB curriculum will aim to empower residents in four competency streams-mental-health maintenance, time management, concise documentation, and effective oral presentation-anchor 14 one-hour Zoom workshops delivered twice weekly over seven weeks (May-June 2025). Each session follows the sequence:

Watch: Pre-assigned 10-minute OME video segment.

Practice: Live case or chart-note exercise in breakout dyads.

Reflect: Group debrief tied to OME-IB strategies

All Zoom calls are recorded; engagement metrics (minutes viewed, etc) are exported via the platform's API for dose-response analyses. Control-arm trainees will receive platform credentials only after the last six-month survey, ensuring contamination is minimized.

Data Acquisition and Quality Control: Surveys are deployed through a HIPAA-compliant REDCap instance with automated email nudges at 48 h and 96 h. De-identified datasets are stored on an encrypted institutional server; access is role-restricted and logged.

Embedded Qualitative Arm At four months into residency, a purposive subsample of intervention participants will undergo 30-45 min semi-structured interviews via Zoom. Using a pragmatic phenomenological lens, will use a mixed inductive/deductive scheme; tri-coder consensus, investigator triangulation, and member-checking will bolster trustworthiness.

ELIGIBILITY:
Inclusion Criteria:

-incoming first year residents

Exclusion Criteria:

* Previous United States accredited postgraduate training
* House Officers
* Physician Assistant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Burnout at 3 months and 6 months. | Baseline measurement, post-intervention measurements at 3 months and 6 months
  The Maslach's burnout inventory is a 22-item measurement of worker burnout which assesses emotional exhaustion (EE), depersonalization (DP), and personal fulfillment (PF) domains. Possible scores range from 0-6 on a Likert scale for each item. Scores oof EE ≥ 27 points, DP ≥ 10, and PF <33 would indicate a high degree of burnout. Scores of EE≤18 points, DP≤5 points, and PF≥40 points would indicate a low degree of burnout.

SECONDARY OUTCOMES:
Change from baseline scores of the CBI-pb subscale at 3 months and 6 months. | Baseline measurement, post-intervention measurements at 3 months and 6 months
  Copenhagen Burnout Inventory personal burnout subscale (CBI-pb) is a tool used to assess personal burnout regardless of the work status.
Mean scores of the Mini ReZ subscales at 6 months | 6-month after the intervention
  The Mini ReZ was adapted from the Mini Z for use in residents, using the Mini Z core 10 questions and 5 additional questions reflecting domains identified by Trockel. The interpretation is based on three subscales: Sub-scale 1 - Supportive Work Environment: add the numbered responses to questions 1-5. Range 5-25 (>=20 is a highly supportive work environment); Sub-scale 2 - Work pace and EHR Stress: add the numbered responses to questions 6-10. Range 5-25 (>=20 is an environment with good pace and manageable EHR stress); Subscale 3 - Resident Experience: add the numbered responses to questions 11-15. Range 5-25 (>=20 is a positive and healthy resident experience).
Proportion of participants whose PHQ-9 total score is ≥ 10 at 3 months and 6 months | Baseline measurement, post-intervention measurements at 3 months and 6 months
  The Patient Health Questionnaire 9-item version (PHQ-9) to assess depressive symptoms. On PHQ-9, depression is categorized as minimal by a score of 0 to 4, mild by a score of 5 to 9, moderate by a score of 10 to 14, moderately severe by a score of 15 to 19, and severe by a score of 20 to 27. A total score ≥ 10 indicates clinically significant depressive symptoms. The outcome is the proportion of participants with a score ≥ 10 at 6 months. Lower proportions reflect better mental-health status.

CONTACTS AND LOCATIONS:
Overall Officials: Raji Ayinla, M.D., CMD, FCCP, FACP, Principal Investigator — New York City Health and Hospitals Corporation
Locations (1):
- Harlem Hospital Center, Manhattan, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the primary and secondary outcome results (baseline demographic variables, intervention allocation, PHQ-9, CBI-PB, EE, Mini-ReZ scores at baseline, 3 months and 6 months, adverse-event indicators) plus the data dictionary and statistical analysis code will be shared. Direct identifiers (name, email, MRN, full dates of birth) and high-risk elements (audio/video files, free-text survey comments) will not be shared to protect confidentiality in this small cohort.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 12 months after publication of the main results and for 5 years via the controlled-access repository Vivli
Access Criteria: Researchers with a methodologically sound proposal, IRB/ethics approval, and a signed data-use agreement may request access through the Vivli platform's review committee.

REFERENCES:
- [Background] Guille C, Zhao Z, Krystal J, Nichols B, Brady K, Sen S. Web-Based Cognitive Behavioral Therapy Intervention for the Prevention of Suicidal Ideation in Medical Interns: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Dec;72(12):1192-8. doi: 10.1001/jamapsychiatry.2015.1880. PMID 26535958
- [Background] Rotenstein LS, Torre M, Ramos MA, Rosales RC, Guille C, Sen S, Mata DA. Prevalence of Burnout Among Physicians: A Systematic Review. JAMA. 2018 Sep 18;320(11):1131-1150. doi: 10.1001/jama.2018.12777. PMID 30326495